CLINICAL TRIAL: NCT05680662
Title: The Study of Quadruple Therapy Quercetin, Zinc, Metformin, and EGCG as Adjuvant Therapy for Early, Metastatic Breast Cancer and Triple-negative Breast Cancer, a Novel Mechanism
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, Dr Amr Ahmed, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amr Ahmed
Record Dates: First submitted 2022-12-23; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer Female; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Quercetin; epigallocatechin gallate; Metformin; Zinc

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- adjuvant quadruple thearpy of quercetin , zinc, EGCG, metformin for 100 breast cancer cases (Experimental): experimental study of adjuvant quadruple therapy of quercetin, zinc, EGCG, and metformin for 100 cases of different types of breast cancer women daily dose as follows daily 500 mg orally quercetin OD daily 50 mg zinc sulfate orally OD daily 300 mg EGCG orally OD daily metformin 850 mg orally OD during chemotherapy courses and until last stage of treatment
  Interventions: Combination Product: quercetin, EGCG, metformin , zinc
- no adjuvant thearpy for 100 cases of breast cancer breast for this group ( controlled group ) (Experimental): this arm ( 100 cases controlled group not taken adjuvant therapy only was taken the regular chemotherapy as prescription
  Interventions: Combination Product: quercetin, EGCG, metformin , zinc

INTERVENTIONS:
Combination Product: quercetin, EGCG, metformin , zinc — this intervention target many mechanisms at tumorigenesis, metastasis autophagy, apoptosis, interleukin 6, cathepsin L, and also epigenetic DNA methylation

SUMMARY:
breast cancer is the most common cancer in women. With more than 1 in 10 new cancer diagnoses each year, It is the second most frequent cancer-related death among women worldwide. Breast cancer develops slowly, and the majority of cases are found through routine screening.

breast cancer-causing deaths among women all over the world and increased in the last few years even though the treatment is advanced like immunotherapy chemotherapy by yet no treatment for triple-negative breast cancer zinc and competition between znt1 and zip6,10 at breast cancer cells. Is zinc ionophore like quercetin and EGCG has a role, In a novel experimental study zinc is a trace metal that has many roles in cells, enzymatic activity, and gene regulations, and also for the integrity of DNA.

Zinc transporters (zinc related -proteins such as ZIPs, and ZnTs are affected by triggers factors like cytokines and growth factors.

There are two large families of zinc transporters like ZIPs ( 14 members) and ZnTs family (10 members), ZIPS family cause an influx of zinc from the extracellular to the cytoplasm and also from intracellular organelles like endoplasmic reticulum or Golgi or mitochondria in contrast to ZnTs which cause an influx of zinc from the cytoplasm to intracellular organelles. ( lower cytoplasmic zinc) (1) Breast cancer deaths occurred from metastasis; Catalytic enzymes called proteases like cathepsin L are frequently overexpressed in aggressive cancers. Breast tumor metastatic potential is correlated with macrophage presence. These macrophages associated with tumors frequently adopt an M2-like pro-tumorigenic phenotype, which results in the production of growth hormones and proteases, notably the lysosomal protease cathepsin L. Because cathepsin L is commonly released by breast cancer cells and aids in tumor invasion, metastasis, and angiogenesis. It is expected that cathepsin L secretion by both tumor-associated macrophages and neoplastic cells would promote the metastatic phenotype because cathepsin L is widely produced by breast cancer cells and helps with tumor invasion, metastasis, and angiogenesis. (2) this study target new mechanisms and achieves the best management as some types of cancer breast like triple-negative breast cancer (TNBC) no definite treatment so we target the following pathways and epigenetic processes by these adjuvant compounds which have a promising role in the immunity like EGCG, Quercetin, Zinc, Metformin so our team will discuss novel methods to achieve the best efficacy from chemotherapy

DETAILED DESCRIPTION:
breast cancer is the most common cancer in women. With more than 1 in 10 new cancer diagnoses each year, It is the second most frequent cancer-related death among women worldwide. Breast cancer develops slowly, and the majority of cases are found through routine screening.

breast cancer-causing deaths among women all over the world and increased in the last few years even though the treatment is advanced like immunotherapy chemotherapy by yet no treatment for triple-negative breast cancer zinc and competition between znt1 and zip6,10 at breast cancer cells. Is zinc ionophore like quercetin and EGCG has a role, In a novel experimental study zinc is a trace metal that has many roles in cells, enzymatic activity, and gene regulations, and also for the integrity of DNA.

Zinc transporters (zinc related -proteins such as ZIPs, and ZnTs are affected by triggers factors like cytokines and growth factors.

There are two large families of zinc transporters like ZIPs ( 14 members) and ZnTs family (10 members), ZIPS family cause an influx of zinc from the extracellular to the cytoplasm and also from intracellular organelles like endoplasmic reticulum or Golgi or mitochondria in contrast to ZnTs which cause an influx of zinc from the cytoplasm to intracellular organelles. ( lower cytoplasmic zinc) (1) Breast cancer deaths occurred from metastasis; Catalytic enzymes called proteases like cathepsin L are frequently overexpressed in aggressive cancers. Breast tumor metastatic potential is correlated with macrophage presence. These macrophages associated with tumors frequently adopt an M2-like pro-tumorigenic phenotype, which results in the production of growth hormones and proteases, notably the lysosomal protease cathepsin L. Because cathepsin L is commonly released by breast cancer cells and aids in tumor invasion, metastasis, and angiogenesis. It is expected that cathepsin L secretion by both tumor-associated macrophages and neoplastic cells would promote the metastatic phenotype because cathepsin L is widely produced by breast cancer cells and helps with tumor invasion, metastasis, and angiogenesis. (2) this study target new mechanisms and achieves the best management as some types of cancer breast like triple-negative breast cancer (TNBC) no definite treatment so we target the following pathways and epigenetic processes by these adjuvant compounds which have a promising role in the immunity like EGCG, Quercetin, Zinc, Metformin so our team will discuss novel methods to achieve the best efficacy from chemotherapy the study will include 100 cases with many types of breast cancer like hormonal sensitive, triple negative, and metastatic breast cancer, and another group of 100 patients not given this adjuvant therapy type of study is a randomized clinical control trial interventional with 4 compounds (EGCG,ZINC, QUERCETIN,METFORMIN)

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18
2. Female patients
3. with any type of breast cancer Ductal carcinoma in situ (DCIS) ... Invasive breast cancer (ILC or IDC) ... Triple-negative breast cancer. ... Inflammatory breast cancer. ... Paget disease of the breast. ... Angiosarcoma. ... Phyllodes tumor.
4. HER2-positive by ASCO CAP 2018 guidelines, confirmed by central testing
5. Participants must have normal organ and marrow function as defined below:

ANC ≥ 1000/mm3 hemoglobin ≥8 g/dl platelets ≥ 75,000/mm3 AST and ALT both <5x institutional ULN Total bilirubin ≤ 1.5 mg/dL. For patients with Gilbert syndrome, the direct bilirubin should be <institutional ULN Serum creatinine ≤ 2.0 mg/dL OR calculated GFR ≥ 30mL/min 6- Locally advanced tumors at diagnosis, including tumors fixed to the chest wall, peau d'orange, skin ulcerations/nodules, or clinical inflammatory changes (diffuse brawny cutaneous induration with an erysipeloid edge) Patients with a history of previous invasive breast cancer.

-

Exclusion Criteria:

Neoadjuvant or adjuvant chemotherapy for this breast cancer prior to enrollment is prohibited.

Any of the following due to teratogenic potential of the study drugs:

Pregnant women Nursing women Women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragms, IUDS, surgical sterilization, abstinence, etc). Hormonal birth control methods are not permitted.

Participants who are receiving any other investigational agents for treatment of breast cancer, unless specific approval is obtained from the Sponsor-Investigator.

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
invasive Disease Free Survival at 3 Years from the time of randomization until the occurrence of the first of the following events: invasive local/regional recurrence, Contralateral invasive breast cancer, Distant recurrence, Death from any cause | Time Frame: 3 Years
  Kaplan-Meier estimates of iDFS will be estimated and plotted with the corresponding 95% confidence intervals.
  from the time of randomization until the occurrence of the first of the following events: invasive local/regional recurrence, Contralateral invasive breast cancer, Distant recurrence, Death from any cause

SECONDARY OUTCOMES:
Invasive Disease Free Survival at 10 Years | 10 years
  Kaplan-Meier estimates of iDFS will be estimated and plotted with the corresponding 95% confidence intervals.
  from the time of randomization until the occurrence of the first of the following events: invasive local/regional recurrence, Contralateral invasive breast cancer, Distant recurrence, Death from any cause
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 [ | 5 years
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting
Total patient chair time of drug administration | 18 months
  Mean difference will be estimated between HP FDC SC and IV admin of HP in sub-study
Breast cancer-specific survival (BCSS) at 10 Years | 10 years
  the time period between randomization and death due to breast cancer.

IPD SHARING:
Plan to Share IPD: Undecided